CLINICAL TRIAL: NCT00222248
Title: The Effect of Pelvic Floor Muscle Training for the Management of Incontinence in Older Women: a Single Blind Randomised Controlled Trial.
Brief Title: Pelvic Floor Muscle Training for Incontinence in Older Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Responsible Party: Principal Investigator, Mary Galea, Professor, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 251632
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Stress Urinary Incontinence
Keywords: Stress urinary incontinence; Pelvic floor muscle training; Bladder training; Older women
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Pelvic floor muscle training (Experimental): Weekly group session of education and exercise to music incorporating pelvic floor muscle training incorporating motor control, strength, endurance, power and functional training in a variety of different positions.
  Interventions: Behavioral: Pelvic floor muscle training and bladder training
- Bladder training (Active Comparator): Weekly group session of education regarding deferral techniques, timed voiding parameters and gentle exercise to music.
  Interventions: Behavioral: Pelvic floor muscle training and bladder training

INTERVENTIONS:
Behavioral: Pelvic floor muscle training and bladder training

SUMMARY:
To determine the effect of pelvic floor muscle training in women aged 70 years and over, who have proven stress urinary incontinence. The hypotheses to be tested are:

1. That pelvic floor muscle training is effective in relief of symptoms of stress urinary incontinence as measured by a greater reduction in the number of episodes of incontinence, quantity of urine lost and improvement of quality of life.
2. That women who undertake pelvic floor muscle training will show greater improvement of pelvic floor muscle function than women who have behavioural (bladder) training, as measured by real time transabdominal ultrasound.

DETAILED DESCRIPTION:
Urinary incontinence is associated with significant personal stress, shame and social stigma and affects around one-third of women over 60 years of age. It restricts the amount of physical activity and can lead to social isolation and poor health. Pelvic floor muscle re-education by physiotherapists is the most commonly recommended method of conservative management. Although a recent Cochrane review concluded that it was an effective treatment for women with stress and mixed incontinence, there is still no strong evidence for the effectiveness of this intervention in elderly women. It has also been suggested that bladder training alone is equally effective in patients with stress urinary incontinence, urge and mixed incontinence. This is contrary to current clinical experience. It is therefore important to distinguish the relative effectiveness of these interventions used in isolation in order to ensure that urinary incontinence is managed in the most effective and efficient way.

Comparisons: pelvic floor muscle training group and bladder training.

Assessments will be conducted at baseline, 1 month, 3 months and 5 months during the intervention period. Both groups will then continue with their home program for a further 7 months until their final assessment (Assessment 5).

Outcome measures will include: volume of urine lost during a stress test, completion of accident diaries, Degree of 'bother', quality of life using the Kings Health Questionnaire, and assessment of pelvic floor function using real time transabdominal diagnostic ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling women aged over 65 years
* urodynamically proven stress incontinence
* Medically stable

Exclusion Criteria:

* Already receiving physiotherapy intervention
* Neurogenic incontinence
* Cannot comply with training program

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 83 (Actual)
Dates: Start 2003-03-03 (Actual); Primary Completion 2006-03-06 (Actual); Study Completion 2006-03-06 (Actual)

PRIMARY OUTCOMES:
Quantity of urine lost over a 7-day period measured by self-report. | 1, 3, 5 (end of intervention) and 12 months
  Self report of urine leakage
Urine lost on stress test measured by pad weigh test. | 1, 3, 5 (end of intervention) and 12 months
  Pad weight following stress test

SECONDARY OUTCOMES:
King's Health Questionnaire. | 1, 3, 5 (end of intervention) and 12 months
  Quality of life questionnaire
Degree of bother | 1, 3, 5 (end of intervention) and 12 months
  Visual Analogue Scale of degree of bother
Severity of stress incontinence | 1, 3, 5 (end of intervention) and 12 months
  Severity of stress incontinence measured by the ICIQ-UI SF
Displacement of pelvic floor during muscle contraction | 1, 3, 5 (end of intervention) and 12 months
  Displacement measured using transabdominal ultrasound imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Mary P Galea, PhD, Principal Investigator — University of Melbourne
Locations (1):
- Austin Health, Melbourne, Victoria, Australia

REFERENCES:
- [Result] Sherburn M, Bird M, Carey M, Bo K, Galea MP. Incontinence improves in older women after intensive pelvic floor muscle training: an assessor-blinded randomized controlled trial. Neurourol Urodyn. 2011 Mar;30(3):317-24. doi: 10.1002/nau.20968. Epub 2011 Jan 31. PMID 21284022